CLINICAL TRIAL: NCT00075920
Title: Technical Development of Strain Rate Echocardiography
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040082; 04-H-0082
Record Dates: First submitted 2004-01-11; First posted 2004-01-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-17

CONDITIONS: Echocardiography, Doppler
Keywords: Heart; Function; Ultrasound; MRI; Left Ventricle; Healthy Volunteer; HV; Heart Disease
MeSH Terms: conditions — Heart Diseases

SUMMARY:
This study will examine heart function using two imaging techniques - echocardiography (ultrasound) and magnetic resonance imaging (MRI) - to evaluate newly developed software for echocardiograph machines. MRI and ultrasound both provide images of the heart structure and function. MRI uses a magnetic field and radio waves to obtain the pictures, while echocardiography uses sound waves.

Patients with any form of heart disease and healthy volunteers 21 years of age and older may be eligible for this study. Candidates must be and able to undergo magnetic resonance imaging and must not have an irregular heart rhythm, heart valve disease, a pacemaker, defibrillator implant, insulin pump, or other metallic implant.

Participants will have two ultrasound examinations and two magnetic resonance imaging examinations, as described below. All the tests will be completed within 24 to 48 hours.

Echocardiography :

For this test, a small probe is passed over the chest. Sound waves emitted from the probe bounce off the heart and are beamed back into the echo machine where they are recorded. The sonographer does a baseline test, which is evaluated by the physician. Then, after a 10- to 20-minute break, portions of the test are repeated. The entire exam takes about 2 hours.

Magnetic Resonance Imaging:

For MRI, the subject lies on a table that slides into a long doughnut-shaped scanner. A small tube is placed in a vein in the hand or arm to give fluids and to infuse gadolinium, a contrast material that brightens the images. Heart rate and blood pressure are monitored during the study, which takes about 3 hours.

DETAILED DESCRIPTION:
The purpose of this protocol is to study the reproducibility of strain rate (SR) echocardiography in normal volunteers and patients with cardiovascular disease. Tissue Doppler ultrasound is a technology which has been validated for the analysis of global and regional left ventricular function and strain and SR measurements are derived from tissue Doppler imaging (TDI) data. Over the last few years, several improvements in echo machine hardware and software have facilitated the rapid acquisition and analysis of tissue Doppler data, and therefore, strain and strain rate information has become easily accessible. Recent publications have demonstrated the usefulness of these techniques in the analysis of systolic and diastolic function of the left ventricle, and in the detection of regional wall motion and ischemia. Several protocols recently initiated in the Cardiovascular Branch involve echocardiographic imaging and include applications of TDI as their primary or secondary endpoints. Therefore, the purpose of this protocol is to allow development of standardized acquisition and analysis methods of TDI for our cardiology protocols and to evaluate the reproducibility of TDI, SR, and strain measurements.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults older than 18 years will be recruited for the CAD group. Since regional wall motion abnormalities, coronary artery disease, and heart failure are rare in subjects under 21, we will limit this group to adults only.

Adults older than age 18 who have undergone surgical repair of Tetralogy of Fallot will be recruited. Normal controls will be age-matched to this group of patients.

Able to provide written informed consent.

EXCLUSION CRITERIA:

Patients with pulmonary artery shunts placed within the last 6 months are not eligible to undergo MRI scanning.

Pregnant or lactating (patients with uncertain pregnancy status will be required to have a screening urine or blood pregnancy test).

Chronic atrial fibrillation; frequent PVC's (more than 1 every 10 heart beats).

Cardiac pacemaker, defibrillator, or other metallic implant which would exclude subject from MRI examination (examples: central nervous system aneurysm clips, implanted neural stimulator, cochlear implant, ocular foreign body, insulin pump, metal shrapnel or bullet).

Inability to provide written informed consent.

Patients with hemoglobinopathies or renal disease with a creatinine clearance (CrCl) less than 20 ml/min will be excluded from MRI sequences involving administration of MRI contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2004-01-08; Study Completion 2007-10-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Katz WE, Gulati VK, Mahler CM, Gorcsan J 3rd. Quantitative evaluation of the segmental left ventricular response to dobutamine stress by tissue Doppler echocardiography. Am J Cardiol. 1997 Apr 15;79(8):1036-42. doi: 10.1016/s0002-9149(97)00043-x. PMID 9114760